CLINICAL TRIAL: NCT01930279
Title: Effect of Sleep Deprivation on Expression of T Cell Markers in Peripheral Blood of Medical Residents
Brief Title: Effect of Partial Sleep Deprivation on Immunological System in Peripheral Blood
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, ayman abu rmaileh, MD, Hadassah Medical Organization
Other Study IDs: LDB001
Record Dates: First submitted 2013-08-25; First posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Sleep Deprivation
Keywords: T cell markers
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- surface markers on T cells as assessed by FACS
  Interventions: Other: Blood withdrawal

INTERVENTIONS:
Other: Blood withdrawal — Blood withdrawal

SUMMARY:
Sleep deprivation was found to affect many organs including the immune system and predisposing for various health consequences including diabetes hypertension infections and increase in neoplastic diseases.

Subjects will be evaluated for immune parameters in peripheral blood test following a regular nigh sleep and compared with a test performed following a night shift in which they slept less than 3 hours.

Each participant will serve as its own control.

DETAILED DESCRIPTION:
Overall Study Design and Plan

1. Subjects will be bled on the day of the experiment between 8and 9 AM.
2. Blood tubes will be tested for T cell markers, serum cytokines levels, and other immune parameters by western blots.
3. The first tube will be tested on the day of experiment.
4. The second tube will kept in the lab and will be tested 24 hours later.
5. The third tube will be kept in the pocket of the subject and be tested 24 hours later.
6. The fourth tube will be kept in the pocket of another subject and will be tested 24 hours later.
7. The subject will be tested again following 24 hours.
8. Each subject will be tested twice following a regular 6-8 hours of sleep, and following an on call duty in which he slept less than 3 hours.

ELIGIBILITY:
Inclusion Criteria:

Male and female ages 18-40 signed confirmed consent no evidence of chronic disease or chronic medications

Exclusion Criteria:

Any type of acute infection or other acute illness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical residnets
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
surface markers of T cell as assessed by FACS | 6 months
serum cytokine levels | 6 months
immune parameters to be assessed by western including STAT proteins | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Jerusalem, Israel